CLINICAL TRIAL: NCT03270774
Title: Central Venous Catheter Colonisation: Prevalence and Associated Factors Among Critically Ill Patients Admitted to Ugandan Intensive Care Units
Brief Title: Central Venous Catheter Colonisation Among Critically Ill Patients in Intensive Care Units
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: CVC Study
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Sepsis; Septic Shock; Post-cardiac Surgery; Post-Cardiorespiratory Arrest Coma; Head Injury; Hypoxic Brain Damage; Acute Liver Failure; Diabetic Ketoacidotic Hyperglycaemic Coma
MeSH Terms: conditions — Sepsis; Shock, Septic; Craniocerebral Trauma; Hypoxia, Brain; Liver Failure, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Central Venous catheter insertion technique and indwelling time are major risk factors for CVC colonisation. Colonisation occurs through microbial migration and biofilm formation along the catheter insertion tract. This study set out to determine the prevalence and associated factors for central venous catheter colonisation among critically ill patient. No data exists in this clinical setting addressing this topic.

Methods: The study population included 100 participants with central venous catheters in situ for at least 24 hours. Catheter tip (distal 5-cm segment) and blood cultures (10mls peripheral blood) were obtained at the time of catheter removal.

DETAILED DESCRIPTION:
Introduction : Central venous catheter (CVC) insertion technique and time spent in situ (dwell period) are major risk factors for CVC colonisation among patients admitted to intensive care units (ICU) worldwide. Normal skin flora colonizes CVCs early in their dwell period (< 7-10 days) causing variable occurrence of infections in all categories of patients. Uganda has no data on CVC colonisation and with increasing use there is concern of CVC colonisation and its consequences. This study was done to determine the prevalence and associated factors of CVC colonization among patients in general ICUs.

Methodology: This was prospective cohort study. Critically ill patients with CVCs in situ from four general ICUs were consecutively enrolled into the study. Data on socio-demographic, clinical characteristics (diagnosis, comorbidities) and CVC insertion (site, technique, experience) was collected using a standardised questionnaire until a sample size of 100 was achieved. At the time of CVC removal, the CVC tip (distal 5cm segment) was aseptically obtained and cultured for microorganisms using the semi-quantitative method. A blood culture sample (10mls) was also collected from a peripheral site at the same time. Data was double entered into EPIDATA version 3.1.5 and exported to STATA version 12.0 for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all age groups were included in this study
* All critically ill patients admitted to the ICU with Central Venous Catheters in situ
* Written informed consent/assent
* Waiver of consent for unconscious patients with no attendant/valid surrogate respondent to provide the required information

Exclusion Criteria:

•Patients who were already on treatment for CVC-related infectious complications.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population All the critically ill patients with CVCs admitted to the general ICUs in the 4 hospitals above during the study period and who met the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Prevalence of central venous catheter colonisation | up to 14 days
  Of the patients that had central venous catheter inserted, how many of them developed central venous catheter colonisation

SECONDARY OUTCOMES:
Prevalence of Central venous catheter associated bloodstream infections | Up to 48 hours after removal of central venous catheter
  Of the patients that developed central venous catheter colonisation, how many of them developed associated bloodstream infection
Factors associated with central venous catheter colonisation | up to 14 days
  Factors that have a significant p-value < 0.5 of association with central venous catheter colonisation